CLINICAL TRIAL: NCT03238807
Title: Effect of Intrauterine Injection of Human Chorionic Gonadotropin Before Embryo Transfer on Clinical Outcomes in In-vitro Fertilization/Intracytoplasmic Sperm Injection Cycles: a Randomized Controlled Trial
Brief Title: Effect of Intrauterine Injection of Hcg Before ET on Clinical Outcomes in IVF/ICSI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Abdallah, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IntraUterine HCG Assiut
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Infertility; ART
Keywords: hCG; Intrauterine hCG; IVF; ICSI
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Group that will receive intrauterine injection of human Chorionic Gonadotropin before ET
  Interventions: Drug: Human Chorionic Gonadotropin
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Drug: Human Chorionic Gonadotropin — 500 IU of human Chorionic Gonadotropin
  Other Names: Epifasi
  Arms: Intervention Group

SUMMARY:
Subfertility is the inability to conceive after 12 months of regular unprotected sexual intercourse. Around 15% of couples suffer from subfertility. As a treatment for subfertility, Assisted Reproductive Techniques (ART) have been a choice for subfertile couples. In Egypt in 2010, Pregnancy Rate was calculated to be 36.2%, Live Birth Rate to be 25.7%.

Implantation is the process by which the embryo adheres to the wall of the uterus. Endometrial receptivity plays the most important role for successful implantation after embryo quality. It is estimated that up to 70% of early pregnancy losses are due to failure of implantation.

Despite extensive research, the embryo-maternal dialogue that orchestrates the implantation process is still not fully understood. Much effort has been done in the last decades to detect factors affecting Implantation and improve endometrial receptivity.

Human Chorionic Gonadotropin (hCG) is a placental glycoprotein hormone that required to maintain pregnancy. Recent research data demonstrates that hCG is secreted very early by the embryo before implantation to facilitate it. hCG has been proved to cause attraction of inflammatory cells, promote angiogenesis, regulate chemical mediators at the endometrium. These effects proceed the classical role of hCG during pregnancy and could be a directly involved in and facilitating the implantation process.

Studies have been conducted to study the effect of injection of different concentrations of hCG inside the uterine cavity before Embryo Transfer (ET) to improve endometrial receptivity and outcomes of In-Vitro Fertilization (IVF) or Intra-Cytoplasmic Sperm Injection (ICSI) cycles.

A recent systematic review was conducted on 12 studies performing intrauterine injection of different doses of hCG before ET. Results of this study showed that there is increased pregnancy outcome after injection of intrauterine 500 IU of hCG. The study recommended a definitive large clinical trial with live birth as the primary outcome. There was no evidence that miscarriage was influenced by intrauterine hCG administration, irrespective of embryo stage at transfer or dose of intrauterine hCG.

Aim of the study:

To detect whether intrauterine injection of hCG before ET improves clinical outcomes in IVF/ICSI cycles.

DETAILED DESCRIPTION:
This study is a Randomized Controlled Trial (RCT) to be done at ART center of Women's Health Hospital, Assiut university, Egypt.

All steps for IVF/ICSI procedure, from the beginning of the induction for controlled ovarian stimulation until just before the procedure of ET, will be done for all enrolled patients as routinely decided according to the local protocol of the ART center in Women Health Hospital, Assiut University. In the day of ET, number and quality of Embryos will be decided according to the routine practice guided by the local protocol.

The intervention preparation will be prepared by adding one vial of hCG containing 5000 IU to 1mL of tissue culture medium (Continuous Single Culture, IrvineScientific). To obtain 500 IU of hCG, 0.1 milliLiter (mL) of the preparation will be injected inside the uterus before ET in the study group. For the control group, 0.1 mL of the tissue culture medium without hCG will be injected inside the uterus before the ET. For both groups we will use Intra-Uterine Insemination (IUI) catheter (Sperm Trans, Sperm Processor) to inject the solution inside the uterine cavity 4 minutes before ET.

We will standardize the procedure of ET for all women apart from the intervention versus control step. All women participating in the study will be put in lithotomy position. Cusco's speculum will be introduced to visualize the cervix. Guided by transabdominal ultrasound with a full bladder, the ET catheter (Cook Sydney IVF Catheter) will be introduced through the cervical os into the uterine cavity. After introduction of the catheter into the uterine cavity loaded embryos will be injected inside the cavity 0.5 cm from the fundus.

Biochemical pregnancy test will be done 14 days after ET by measuring hCG in the woman's serum. If the test result is positive (according to the standard values that is used in the laboratory), a transvaginal ultrasound will be done 3 weeks following the positive biochemical test, to document the visualization of gestational sac, fetal pole and cardiac pulsation.

Pregnancy rate (PR) is calculated by the number of women with positive biochemical pregnancy test to the number of women enrolled in each group. The clinical pregnancy was defined as a viable pregnancy when there is evidence of a gestational sac, embryo and fetal heart rate at the time of ultrasound evaluation. Clinical Pregnancy Rate (cPR) is calculated by the percentage of detected clinical pregnancies using ultrasound to the IVF/ICSI cycles in each group. Implantation rate (IR) is calculated by the number of visualized embryos by transvaginal ultrasound to the number of transferred embryos. While Live Birth Rate (LBR) is calculated by the number of live births to the number of transferred embryos. Miscarriage rate (MR) is calculated by the ratio of miscarriages to the number of confirmed pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* infertility, male or female factor
* Women undergoing ICSI/IVF

Exclusion Criteria:

* functional azoospermia
* submucous uterine myomas or previous myomectomy
* endometriosis
* hydrosalpinges without prior excision or occlusion of the tubal ostia

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2020-10-04 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate (LBR) | 9 months
  calculated by the number of live births to the number of transferred embryos

SECONDARY OUTCOMES:
Clinical Pregnancy Rate (cPR) | 5 weeks
  calculated by the percentage of detected clinical pregnancies using ultrasound to the IVF/ICSI cycles in each group
Implantation Rate (IR) | 5 weeks
  calculated by the number of visualized embryos by transvaginal ultrasound to the number of transferred embryos
Miscarriage rate (MR) | 3 months
  calculated by the ratio of miscarriages to the number of confirmed pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Makhlouf, MD, Principal Investigator — Assiut University; Hazem Saadeldine, MD, Study Chair — Assiut University; Esraa Badran, MD, Study Chair — Assiut University; Karim Abdallah, M.Sc, Study Director — Assiut University
Locations (1):
- Assiut University - Women's Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification to Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately after publication indefinitely.
Access Criteria: Proposals should be directed to karimsayed88@hotmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Abdallah KS, Makhlouf A, Badran E, El-Nashar IM, Al-Hussaini TK, Farghaly T, Mohamed HS, Mol BW, Abdelmagied AM. Intrauterine injection of HCG before embryo transfer: a parallel, double-blind randomized trial. Reprod Biomed Online. 2021 Oct;43(4):663-669. doi: 10.1016/j.rbmo.2021.06.011. Epub 2021 Jun 20. PMID 34412973